CLINICAL TRIAL: NCT05020990
Title: The Comparative Clinical Performance of Two Daily Disposable Toric Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: C20-691 (EX-MKTG-121)
Record Dates: First submitted 2021-08-19; First posted 2021-08-25 (Actual); Results first posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-09

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Lens A, then Lens B (Experimental): Participants wore Lens A for one week, then crossed over to wear Lens B for one week.
  Interventions: Device: Lens A (delefilcon A); Device: Lens B (stenfilcon A)
- Lens B, then Lens A (Experimental): Participants wore Lens B for one week, then crossed over to wear Lens A for one week.
  Interventions: Device: Lens A (delefilcon A); Device: Lens B (stenfilcon A)

INTERVENTIONS:
Device: Lens A (delefilcon A) — Daily disposable for one week
Device: Lens B (stenfilcon A) — Daily disposable for one week

SUMMARY:
This study aimed to compare the clinical performance of two daily disposable toric contact lenses.

DETAILED DESCRIPTION:
This was a multi-center, randomized, participant-masked, bilateral study controlled by cross-comparison. Participants were assigned to either lens type in random sequence. Lenses were worn on a daily disposable wear schedule. Follow-up visits for each lens were performed after 1 week of wear.

ELIGIBILITY:
Inclusion Criteria:

1. They are at least 18 years old and have the capacity to volunteer.
2. They understand their rights as a research subject and are willing and able to sign a Statement of Informed Consent.
3. They are willing and able to follow the protocol.
4. They currently wear soft contact lenses or have done so in the past two years.
5. They have a spherical component of their contact lens prescription between Plano to - 6.00DS (inclusive).
6. They have a cylindrical component of their contact lens prescription between -0.75DC and -2.50DC (inclusive).
7. They can be satisfactorily fitted with the study lens types.
8. At dispensing, they could attain at least 0.20 logMAR distance high contrast visual acuity in each eye with the study lenses within the available power range.
9. They are willing to comply with the wear schedule (at least five days per week and for at least eight hours per day).
10. They own a wearable pair of spectacles.
11. They agree not to participate in other clinical research while enrolled on this study.

Exclusion Criteria:

1. They have an ocular disorder which would normally contra-indicate contact lens wear.
2. They have a systemic disorder, which would normally contra-indicate contact lens wear.
3. They are using any topical medication such as eye drops or ointment.
4. They are aphakic.
5. They have had corneal refractive surgery.
6. They have any corneal distortion resulting from previous hard or rigid lens wear or have keratoconus.
7. They are pregnant or breastfeeding.
8. They have any ocular abnormality which would, in the opinion of the investigator, normally contraindicate contact lens wear.
9. They have eye or health conditions including immunosuppressive or infectious diseases, which would, in the opinion of the investigator, contraindicate contact lens wear or pose a risk to study personnel; or a history of anaphylaxis or severe allergic reaction.
10. They are currently wearing one of the study contact lenses.
11. They have taken part in any other contact lens or care solution clinical trial or research, within two weeks prior to starting this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Morgan, Principal Investigator — Eurolens Research
Locations (3):
- United Kingdom (3):
  - Cameron Optometry, Edinburgh, Edinburg
  - Simon Falk Eyecare, Oakwood, Leeds
  - Phipps Opticians, Heckmondwike

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 55 participants were dispensed study lenses, and 54 completed the study. Five participants discontinued the study prior to dispensing and were therefore not included in either the enrollment count or data analysis population. Nine participants were ineligible.
Pre-assignment Details: Five participants were initially ineligible, but were re-enrolled following a protocol amendment that expanded the age range and allowed the use of an increased range of lens axes for Lens A.
Groups:
- Lens A (Delefilcon A), Then Lens B (Stenfilcon A): Participants wore Lens A for one week, then crossed over to wear Lens B for one week.
- Lens B (Stenfilcon A), Then Lens A (Delefilcon A): Participants wore Lens B for one week, then crossed over to wear Lens A for one week.
Period: Period 1 (One Week)
Arm/Group | Lens A (Delefilcon A), Then Lens B (Stenfilcon A) | Lens B (Stenfilcon A), Then Lens A (Delefilcon A)
Started | 28 | 26
Completed | 28 | 26
Not Completed | 0 | 0
Period: Period 2 (One Week)
Arm/Group | Lens A (Delefilcon A), Then Lens B (Stenfilcon A) | Lens B (Stenfilcon A), Then Lens A (Delefilcon A)
Started | 28 | 26
Completed | 28 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: All participants who were dispensed lenses and successfully completed the study.
Arm/Group | Overall Study
Number analyzed (Participants) | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.6 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Subjective Handling Rating on Lens Removal
Description: Subjective handling rating on lens removal was measured on a scale of 0-100 where 0=Unmanageable and 100=Excellent removal.
Time Frame: One week
Population: Lens A: all data for one participant was discounted, as the follow-up visit took place significantly outside the date range for this visit.
  Lens B: all data for a different participant was discounted, as the follow-up visit took place significantly outside the date range for this visit. Another participant's subjective scores and symptoms were not collected at the correct study visit in error, and their data was subsequently excluded from analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Lens A: Participants that received Lens A during either the first or second period of the study.
- Lens B: Participants that received Lens B during either the first or second period of the study.
Arm/Group | Lens A | Lens B
Number analyzed (Participants) | 53 | 52
units on a scale | 85.5 (17.7) | 83.3 (20.1)

2. Secondary Outcome: Overall Lens Fit at Follow-up
Description: Lens fit was reported as either optimum, acceptable, or unacceptable. To determine this, lens fit parameters (horizontal centration, vertical centration, corneal coverage, and lens movement) were measured on a 5-point scale (-2 to +2), where -2=Extremely nasal, 0=Optimum, and +2=Extremely temporal. Scores between -1 and +1 were considered "Acceptable". For overall lens fit to be 'acceptable', no parameters could be extreme. For a score to be 'optimum', all parameters needed to be optimum.
Time Frame: One Week
Population: Lens A: all data for one participant was discounted, as the follow-up visit took place significantly outside the date range for this visit.
  Lens B: all data for a different participant was discounted, as the follow-up visit took place significantly outside the date range for this visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Lens A | Lens B
Number analyzed (Participants) | 53 | 53
Participants
  Optimum | 23 | 20
  Acceptable | 53 | 53
  Unacceptable | 0 | 0

3. Secondary Outcome: Biomicroscopy Score at Follow-up
Description: Slit lamp biomicroscopy was used to assign grades to various biomicroscopic signs, as assessed by investigator, using Efron Grading Scales scored to the nearest 0.1 unit. Grading ranged from 0-4, where 0=None and 4=Severe.
Time Frame: One week
Population: Lens A: all data for one participant was discounted, as the follow-up visit took place significantly outside the date range for this visit.
  Lens B: all data for a different participant was discounted, as the follow-up visit took place significantly outside the date range for this visit. For parameter 'mucin balls', data from an additional participant was not collected in error.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lens A | Lens B
Number analyzed (Participants) | 53 | 53
score on a scale
  Limbal hyperaemia | 0.63 (0.41) | 0.64 (0.40)
  Conjunctival hyperaemia | 0.82 (0.32) | 0.76 (0.31)
  Corneal vascularisation | 0.05 (0.15) | 0.03 (0.09)
  Corneal oedema | 0.00 (0.00) | 0.00 (0.00)
  Corneal staining | 0.23 (0.37) | 0.20 (0.32)
  Conjunctival staining | 0.41 (0.44) | 0.53 (0.49)
  Papillary conjunctivitis | 0.90 (0.40) | 0.90 (0.43)
  Blepharitis | 0.06 (0.16) | 0.06 (0.15)
  Meibomian gland dysfunction | 0.16 (0.32) | 0.09 (0.18)
  Mucin balls: number analyzed (Participants) | 53 | 52
  Mucin balls | 0.00 (0.00) | 0.10 (0.69)

ADVERSE EVENTS:
Time Frame: The duration of the study, approximately 2 weeks per participant.
Description: There was 1 significant ocular adverse event and 1 non-significant ocular adverse event in 2 separate participants that occurred while wearing their habitual lens.
Arm/Group | Lens A | Lens B
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/54
Other Adverse Events (participants affected / at risk) | 5/54 | 1/54
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lens A (N=54) | Lens B (N=54)
Swelling of Eyelid (Eye disorders) | 0 (0) | 1 (1)
Eye Redness (Eye disorders) | 1 (1) | 0 (0)
Corneal Scar (Eye disorders) | 1 (1) | 0 (0)
Corneal Abrasion (Eye disorders) | 1 (1) | 0 (0)
Conjunctival Redness (Eye disorders) | 2 (2) | 0 (0) — Possibly due to mechanical irritation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-03): https://cdn.clinicaltrials.gov/large-docs/90/NCT05020990/Prot_SAP_000.pdf